CLINICAL TRIAL: NCT05626296
Title: Molecular Network Characteristics of Phlegm-heat Syndrome in Ischemic Stroke Based on Multi-omics Integrated Analysis
Status: Recruiting | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Other Study IDs: 82102823-01
Record Dates: First submitted 2022-11-14; First posted 2022-11-23 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phlegm-heat syndrome in ischemic stroke: Phlegm-heat syndrome: the score of "Phlegm-dampness syndrome" ≥10 with the score of "Internal fire syndrome" ≥10 in Diagnostic Scale for Syndrome Elements of Ischemic Stroke
- Non-phlegm-heat syndrome in ischemic stroke: Non-phlegm-heat syndrome: the score of "Phlegm-dampness syndrome" <10 with the score of "Internal fire syndrome" <10 in Diagnostic Scale for Syndrome Elements of Ischemic Stroke
- Healthy subjects

SUMMARY:
The molecular characteristics of ischemic stroke with phlegm-heat syndrome and candidate biomarkers were identified based on multi-omics data. The main purpose of this study is to validate the molecular characteristics and biomarkers of phlegm-heat syndrome in ischemic stroke, and to demonstrate the association of biomarkers with clinical outcomes.

DETAILED DESCRIPTION:
This is a cohort study in patients with ischemic stroke. The demographic characteristics, TCM syndromes, and other baseline information will be recorded. At the same time, baseline peripheral blood will be collected. These participants will be followed up to 90 days of onset, and 90-day modified Rankin scale (mRS) scores will be assessed. The collected blood samples will be tested by multi-factor detection technology for candidate biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke, were confirmed by magnetic resonance imaging (MRI).
* Symptom onset within 72 hours.
* Diagnosis of phlegm-heat syndrome or non-phlegm-heat syndrome.
* Male or female ≥ 50 years and ≤ 80 years.
* With written informed consent.

Exclusion Criteria:

* Planned or already receiving intravenous thrombolysis or endovascular treatment.
* Acute infectious diseases or acute exacerbations of chronic diseases within one month before enrollment.
* Patients with previous stroke.
* Renal or hepatic insufficiency, tumors, immune diseases, severe underlying diseases.
* Other conditions that may affect the collection and evaluation of clinical information (e.g., severe aphasia, mental illness).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 50 to 80 years with acute ischemic stroke within 72 hours of onset. Moreover, these patients fit the diagnosis of phlegm-heat syndrome or non-phlegm-heat syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Omic biomarkers associated with phelm-heat syndrome in ischemic stroke | baseline
  Sensitivity, specificity, and area under the ROC curve of omic biomarkers of Phlegm-heat syndrome in ischemic stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China